CLINICAL TRIAL: NCT00121277
Title: A Phase I Study of Suberoylanilide Hydroxamic Acid (SAHA) in Combination With Capecitabine in Patients With Solid Tumors
Brief Title: Vorinostat and Capecitabine in Treating Patients With Metastatic or Unresectable Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PMH-PHL-035; CDR0000434850 (Registry Identifier: PDQ (Physician Data Query)); NCI-6868
Record Dates: First submitted 2005-07-19; First posted 2005-07-21 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-07

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Capecitabine; Vorinostat

ARMS (1):
- SAHA (Suberoylanilide Acid) with Capecitabine (Experimental)
  Interventions: Drug: capecitabine; Drug: vorinostat

INTERVENTIONS:
Drug: capecitabine
Drug: vorinostat

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as vorinostat and capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Vorinostat may also stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of vorinostat and capecitabine in treating patients with unresectable or metastatic solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose and recommended phase II dose of vorinostat (SAHA) and capecitabine in patients with metastatic or unresectable solid tumors.
* Determine the safety and tolerability of this regimen in these patients.

Secondary

* Correlate the clinical effects with the pharmacokinetic effects of this regimen in these patients.

OUTLINE: This is a dose-escalation, multicenter study.

Patients receive oral vorinostat (SAHA) once or twice daily and oral capecitabine twice daily on days 1-14. Treatment repeats every 21 days for at least 6 courses in the absence of disease progression or unacceptable toxicity. Patients achieving a complete response (CR) receive 2 courses beyond documentation of CR. Patients achieving a partial response receive 2 courses beyond documentation of best response.

Cohorts of 3-6 patients receive escalating doses of SAHA and capecitabine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. An additional 12 patients are treated at the MTD.

After completion of study treatment, patients are followed at 3-4 weeks and then every 3 months thereafter.

PROJECTED ACCRUAL: Approximately 18-30 patients will be accrued for this study within 6-10 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignant solid tumor

  * Metastatic or unresectable disease
* Standard curative or palliative measures do not exist or are no longer effective
* Patients who received prior radiotherapy must have measurable disease outside a previously irradiated field OR disease progression after prior radiotherapy
* No known brain metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2 OR
* Karnofsky 60-100%

Life expectancy

* More than 12 weeks

Hematopoietic

* WBC ≥ 3,000/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* Bilirubin normal
* AST and ALT ≤ 2.5 times upper limit normal (ULN)

Renal

* Creatinine normal OR
* Creatinine clearance ≥ 60 mL/min

Cardiovascular

* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Able to swallow oral medication
* No clinical or radiological diagnosis of bowel obstruction
* No ongoing or active infection
* No history of allergic reaction attributed to compounds of similar chemical or biological composition to suberoylanilide hydroxamic acid or other agents used in this study
* No known dihydropyrimidine dehydrogenase deficiency
* No psychiatric illness or social situation that would preclude study compliance
* No other uncontrolled illness

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered
* Prior fluorouracil allowed
* No prior capecitabine

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics
* More than 4 weeks since prior radiotherapy and recovered
* No prior radiotherapy to > 40% of bone marrow

Surgery

* At least 4 weeks since prior surgery and recovered

Other

* At least 2 weeks since prior valproic acid
* No other concurrent investigational agents
* No other concurrent anticancer therapy
* No concurrent combination antiretroviral therapy for HIV-positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2005-09; Primary Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated doses of vorinostat (SAHA) and capecitabine | 1 cycle
Safety and tolerability as assessed by CTCAE v3.0 | All cycles

SECONDARY OUTCOMES:
Response rate as assessed by RECIST criteria | Every 2 cycles
Molecular markers as assessed by molecular analysis | Cycle 1
Survival | progression free survival every 2 cycles

CONTACTS AND LOCATIONS:
Overall Officials: Eric X. Chen, MD, PhD, Principal Investigator — Princess Margaret Hospital, Canada
Locations (2):
- Canada (2):
  - Ottawa Hospital Regional Cancer Centre - General Campus, Ottawa, Ontario
  - Princess Margaret Hospital, Toronto, Ontario